CLINICAL TRIAL: NCT03285919
Title: Feasibility of Perturbed-balance Training During Treadmill Walking in a High-functioning Chronic Stroke Subject: a Case-control Study
Brief Title: Perturbed-balance Training During Treadmill Walking for Stroke Subjects
Acronym: BALANCESI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: URIS201703
Record Dates: First submitted 2017-09-05; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Stroke
Keywords: perturbed walking; stepping response
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case - stroke survivor (Experimental): Stroke survivor, 6mon post stroke resulting in right-sided hemiparesis, 53yrs old, had completed a 2mon rehabilitation program prior to the study. He underwent 30 training sessions with the Balance Assessment Robot (BAR™) within a 10-week period, each consisting of 10-15min of unperturbed treadmill and 30-45min of perturbation training. Perturbations were delivered in the forward, backward, left and right direction, occurring every 6sec, at the left leg initial contact and the right leg initial contact. Two training sessions were spent to determine adequate treadmill speed (0.4m/s) and perturbation amplitude (60N), followed by the first assessment session. After the last training session, assessment was repeated using the same parameters plus 90N perturbation amplitude.
  Interventions: Device: Balance Assessment Robot (BAR™)
- Control - matched healthy subject (Active Comparator): Healthy male, height- and weight-matched to the Case. He was assessed according to the same protocol as the Case using the Balance Assessment Robot (BAR™) at perturbation amplitudes 60 and 90 N.
  Interventions: Device: Balance Assessment Robot (BAR™)

INTERVENTIONS:
Device: Balance Assessment Robot (BAR™) — The BAR™ has got six degrees of freedom (DOF) that interface to the pelvis of a walking subject. Five DOFs (translation of pelvis in sagittal, lateral and vertical directions; pelvic rotation and pelvic list) are actuated and admittance-controlled, providing transparent haptic interaction with negligible power transfer; the remaining DOF (pelvic tilt) is passive. The BAR™ is capable of delivering perturbations in the directions forward/backward and left/right, but for the purpose of this study only "outward" perturbations in the frontal plane were considered.

SUMMARY:
A control and a post-stroke subject with right-side chronic hemiparesis were studied. The post-stroke subject underwent 30 sessions of balance-perturbed training while walking on an instrumented treadmill where the Balance Assessment Robot (BAR™) randomly delivered pushes to pelvis in various directions at various speeds and at various perturbation amplitudes. The investigators assessed kinematics, kinetics, electromiography and spatio-temporal responses to outward-directed perturbations commencing either at foot contact of the left or the right leg.

DETAILED DESCRIPTION:
For a detailed description of the study, see the Arms and Interventions section.

ELIGIBILITY:
Inclusion criteria:

* Case: community-dwelling, high-functioning stroke survivor
* Control: healthy volunteer, height- and weight-matched to the Case

Exclusion criteria:

* any disease or injury affecting cognition
* any disease or injury affecting balance or gait

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Change in centre of mass of the Case | Assessment at session no. 3 (during week 1) and session no. 30 (during week 10)
  For the purpose of qualitative assessment of kinematics and kinetics
Change in centre of pressure of the Case | Assessment at session no. 3 (during week 1) and session no. 30 (during week 10)
  For the purpose of qualitative assessment of kinematics and kinetics
Change in ground reaction force of the Case | Assessment at session no. 3 (during week 1) and session no. 30 (during week 10)
  For the purpose of qualitative assessment of kinematics and kinetics

SECONDARY OUTCOMES:
Centre of mass of the Control | During the only session (i.e., session 1 on day 1)
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping
Centre of pressure of the Control | During the only session (i.e., session 1 on day 1)
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping
Ground reaction force of the Control | During the only session (i.e., session 1 on day 1)
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping

OTHER OUTCOMES:
Step length | During both assessment sessions for the Case (i.e., session no. 3 during week 1, and session no. 30 during week 10); during the only session (i.e., session 1 on day 1) for the Control
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping
Step width | During both assessment sessions for the Case (i.e., session no. 3 during week 1, and session no. 30 during week 10); during the only session (i.e., session 1 on day 1) for the Control
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping
Step time | During both assessment sessions for the Case (i.e., session no. 3 during week 1, and session no. 30 during week 10); during the only session (i.e., session 1 on day 1) for the Control
  For the purpose of qualitative assessment of spatio-temporal characteristics of stepping
Electromiography (at M. tibialis anterior, M. soleus, M. gastrocnemius lat., M. gastrocnemius med., M. rectus femoris, M. semitendinosus, M. gluteus med., M. gluteus max.) | During both assessment sessions for the Case (i.e., session no. 3 during week 1, and session no. 30 during week 10); during the only session (i.e., session 1 on day 1) for the Control
  For the purpose of qualitative assessment

CONTACTS AND LOCATIONS:
Overall Officials: Zlatko Matjačić, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Olensek A, Zadravec M, Matjacic Z. A novel robot for imposing perturbations during overground walking: mechanism, control and normative stepping responses. J Neuroeng Rehabil. 2016 Jun 11;13(1):55. doi: 10.1186/s12984-016-0160-7. PMID 27287551
- [Derived] Matjacic Z, Zadravec M, Olensek A. Feasibility of robot-based perturbed-balance training during treadmill walking in a high-functioning chronic stroke subject: a case-control study. J Neuroeng Rehabil. 2018 Apr 11;15(1):32. doi: 10.1186/s12984-018-0373-z. PMID 29642921